CLINICAL TRIAL: NCT04946214
Title: A Pilot Study Using a Digital Behavioral Intervention With a Smart Water Bottle to Improve Bladder Filling Compliance in Prostate Cancer Patients Undergoing Radiation Therapy
Brief Title: A Behavioral Health Intervention Using Digital Technology in Radiation Therapy for Prostate Cancer Patients
Acronym: HIDRATEPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Alan Dal Pra, Associate Professor of Clinical Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20200017
Record Dates: First submitted 2021-06-01; First posted 2021-06-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Radiation Toxicity
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart Water Bottle Intervention Arm (Other): Patients will receive a smart water bottle, then instructed on bowel and bladder preparation for daily standard of care radiotherapy treatments for up to 10 weeks.
  Interventions: Behavioral: Smart Water Bottle

INTERVENTIONS:
Behavioral: Smart Water Bottle — Patients will be given a smart water bottle and coached on its use. The device is a 24 oz non-bisphenol A acrylic water bottle with the ability to track water consumption from the bottle, alert its users via a smartphone-based notification system, as well as visually remind patients with a light-emitting diode in the device. Participants will be alerted to drink patient-specific volumes of room temperature water 45 minutes prior to daily standard of care radiotherapy.

SUMMARY:
The purpose of this study is to determine how to incorporate a smart water bottle to improve bladder filling for prostate cancer patients undergoing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 17 but less than 81.
* Non-metastatic prostate cancer patients undergoing definitive radiation treatment.
* Patients that self-identify as "smartphone owners".
* Patients with either iPhone (iOS 13.0 or higher) or Android (version 5.0.1 or higher) based smartphone access.
* English or Spanish speaking patients.

Exclusion Criteria:

* Patients with any history of pre-existing urinary retention.
* Patients with any history of kidney, urothelial tract or bladder cancer.
* Post-operative prostate patients.
* Patients that plan to be treated with pelvic lymph node radiation coverage.
* Patients without a functional bladder.
* Patients with a history of prior pelvic surgery or penile augmentation (circumcision is okay).
* Patients who have previously received any form of pelvic radiation.
* Patients unable to give informed consent.
* Patients who refuse to drink room-temperature water used for bladder filling.
* Patients without functional vision.
* Patients who are colorblind.
* Patient who refuse to use the smartphone app or who refuse consent.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who did not continue to use the intervention through the study. | Up to 10 weeks
  Proportion of participants will be reported as those who did not continue to use the intervention throughout the study.

SECONDARY OUTCOMES:
Proportion of non-compliant participants as measured by survey | Up to 10 weeks
  Proportion of non-compliant participants via a patient-reported survey.
Proportion of non-compliant participants as measured by bladder volume | Up to 10 weeks
  Non-compliance to study intervention will be assessed using a cone beam Computerized Tomography (CT) scan of participant's bladder volume
Bladder volumetric measurements | Up to 10 weeks
  As measured by cone beam CT scan
Rectum Volumetric Measurements | Up to 10 weeks
  As measured by cone beam CT scan
Patient's perception of bladder filling compliance as measured by Service User Technology Acceptability Questionnaire | Up to 10 weeks
  Patient reported scores based on Service User Technology Acceptability Questionnaire (SUTAQ) will measure patient's perception of the smart water bottle. SUTAQ has a total score ranging from 20-100 with the higher score indicating increased user acceptability and comfort with the device.
Proportion of patients refusing participation | Baseline
  Proportion of screen-eligible participants who refused study participation

CONTACTS AND LOCATIONS:
Overall Officials: Alan Dal Pra, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Lennar Medical Foundation, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin W, Montoya C, Rich BJ, Taswell CS, Noy M, Kwon D, Spieler B, Mahal B, Abramowitz M, Yechieli R, Pollack A, Dal Pra A. A Smart Water Bottle and Companion App (HidrateSpark 3) to Improve Bladder-Filling Compliance in Patients With Prostate Cancer Receiving Radiotherapy: Nonrandomized Trial of Feasibility and Acceptability. JMIR Cancer. 2024 Sep 10;10:e51061. doi: 10.2196/51061. PMID 39255484